CLINICAL TRIAL: NCT01282463
Title: An Open-Label, Multicenter, Randomized Phase 2 Study Evaluating the Safety and Efficacy of Docetaxel in Combination With Ramucirumab (IMC-1121B) Drug Product or IMC-18F1 or Without Investigational Therapy as Second-line Therapy in Patients With Locally Advanced or Metastatic Transitional Cell Carcinoma of the Bladder, Urethra, Ureter, or Renal Pelvis Following Disease Progression on First-line Platinum-based Therapy
Brief Title: Study of Ramucirumab or Icrucumab (IMC-18F1) With Docetaxel or Docetaxel Alone as Second-Line Therapy in Participants With Bladder,Urethra, Ureter, or Renal Pelvis Carcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 13943; CP20-0902 (Other: ImClone Systems); I4Y-IE-JCDC (Other: Eli Lilly and Company)
Record Dates: First submitted 2011-01-21; First posted 2011-01-25 (Estimated); Results first posted 2019-07-02 (Actual); Last update posted 2019-09-09 (Actual); Status verified 2019-08

CONDITIONS: Carcinoma of Urinary Tract; Urethral Carcinoma; Carcinoma of Ureter; Carcinoma of Renal Pelvis
Keywords: Carcinoma, Renal Cell
MeSH Terms: conditions — Urethral Neoplasms; Ureteral Neoplasms; Carcinoma, Renal Cell | interventions — Docetaxel; Ramucirumab; Icrucumab; IMC-18F1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Docetaxel (Active Comparator): Cycles repeat every 3 weeks until disease Progression, unacceptable toxicity, or withdrawal.
  Interventions: Drug: Docetaxel
- Docetaxel + Ramucirumab DP (Experimental): Cycles repeat every 3 weeks until disease Progression, unacceptable toxicity, or withdrawal.
  Interventions: Drug: Docetaxel; Biological: Ramucirumab DP
- Docetaxel + Icrucumab (Experimental): Cycles repeat every 3 weeks until disease Progression, unacceptable toxicity, or withdrawal.
  Interventions: Drug: Docetaxel; Biological: Icrucumab

INTERVENTIONS:
Drug: Docetaxel — Docetaxel: 75 milligram/square meter (mg/m2) on Day 1 of each 21-day cycle
Biological: Ramucirumab DP — Ramucirumab (DP): 10 milligram/kilogram (mg/kg) intravenous (IV) on day 1 of each 21-day cycle
  Other Names: IMC-1121B; LY3009806
  Arms: Docetaxel + Ramucirumab DP
Biological: Icrucumab — 12 mg/kg I.V. on day 1 and Day 8 of each 21-day cycle
  Other Names: IMC-18F1; LY3012212
  Arms: Docetaxel + Icrucumab

SUMMARY:
This multicenter trial will enroll participants with metastatic transitional cell carcinoma of the bladder, urethra, ureter, or renal pelvis who have had disease progression on first-line platinum-based chemotherapy regimens. Participants will be enrolled into 1 of 3 treatment arms: docetaxel; docetaxel and ramucirumab; or docetaxel and icrucumab.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed transitional cell carcinoma of the bladder, urethra, ureter, or renal pelvis
* Locally advanced or metastatic and unresectable transitional cell carcinoma of the bladder, urethra, ureter, or renal pelvis
* Had treatment with a platinum-containing regimen
* Disease progression within 12 months of after receiving the last dose of a platinum containing regimen in the neoadjuvant or adjuvant setting, and/or had disease progression while on a platinum-containing regimen or within 12 months after the last dose of therapy in the locally advanced or metastatic setting
* Has measurable or nonmeasurable disease
* Life expectancy of ≥ 3 months
* Received no more than 2 prior systemic chemotherapy regimens in any setting
* Has an Eastern Cooperative Oncology Group (ECOG) performance status of 0-1
* Has adequate hematologic, coagulation, hepatic and renal function
* Does not have:

  * cirrhosis at a level of Child-Pugh B (or worse)
  * cirrhosis (any degree) and a history of hepatic encephalopathy or ascites resulting from cirrhosis and requiring ongoing treatment with diuretics and/or paracentesis
* If female, is surgically sterile, postmenopausal, or compliant with a highly effective contraceptive method during and for 12 weeks after the treatment period
* If male, the patient is surgically sterile or compliant with a contraceptive regimen during and for 12 weeks after the treatment period

Exclusion Criteria:

* Received more than one prior systemic treatment regimen for metastatic disease
* Received prior systemic taxane therapy (except for prior paclitaxel therapy) for Transitional Cell Carcinoma of the bladder, urethra, ureter, or renal pelvis in any setting (neoadjuvant, adjuvant, metastatic). Prior intravesical taxane therapy is allowed
* Has received more than one prior anti-angiogenic agent for Transitional Cell Carcinoma of the bladder, urethra, ureter, or renal pelvis
* Has received radiation therapy within 4 weeks prior to randomization
* Has a history of uncontrolled hereditary or acquired bleeding or thrombotic disorders
* Has experienced a Grade ≥ 3 bleeding event (eg, via gastric ulcers, gastric varices, or gross hematuria) within 3 months prior to randomization
* Has uncontrolled intercurrent illness including, but not limited to symptomatic anemia, uncontrolled hypertension, symptomatic congestive heart failure, unstable angina pectoris, symptomatic or poorly controlled cardiac arrhythmia, psychiatric illness/social situations, or any other serious uncontrolled medical disorders
* Has experienced any arterial thrombotic or thromboembolic events, including but not limited to myocardial infarction, transient ischemic attack or cerebrovascular accident, within 6 months prior to randomization
* Has known brain metastases, uncontrolled spinal cord compression, or leptomeningeal disease
* Has an ongoing or active infection requiring parenteral antibiotic, antifungal, or antiviral therapy
* Has known human immunodeficiency virus infection or acquired immunodeficiency syndrome
* Has received a prior autologous or allogeneic organ or tissue transplantation
* Received chemotherapy within 21 days prior to randomization; and/or is currently enrolled in, or discontinued within 21 days prior to randomization from, a clinical trial involving an investigational product or unapproved use of a drug or device (other than the study drug[s] used in this study), or is concurrently enrolled in any other type of medical research judged not to be scientifically or medically compatible with this study; and/or was treated with anti-angiogenic therapy within 28 days prior to randomization
* Has undergone major surgery within 28 days prior to randomization, or subcutaneous venous access device placement within 7 days prior to randomization
* Has had a serious nonhealing wound, ulcer, or bone fracture within 28 days prior to randomization
* Has an elective or planned major surgery to be performed during the course of the trial
* Is pregnant or lactating
* Has a concurrent active malignancy other than adequately treated non-melanomatous skin cancer, curatively treated cervical carcinoma in-situ, other noninvasive carcinoma or in-situ neoplasm, or prostate cancer with an undetectable prostate specific antigen (PSA) and no current treatment with hormone therapy
* Has an acute/subacute bowel obstruction or history of chronic diarrhea requiring ongoing medical intervention
* History of gastrointestinal perforation and/or fistula within 6 months prior to randomization
* Has active diverticulitis
* Known hypersensitivity to docetaxel or other drugs formulated with polysorbate 80
* Known hypersensitivity to agents of similar biologic composition as ramucirumab DP, IMC-18F1, or other agents that specifically target vascular endothelial growth factor receptor (VEGF)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 148 (Actual)
Dates: Start 2011-04; Primary Completion 2015-02 (Actual); Study Completion 2015-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (32):
- United States (26):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Los Angeles, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Sacramento, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., San Francisco, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Aurora, Colorado
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., New Haven, Connecticut
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Washington D.C., District of Columbia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Boca Raton, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Jacksonville, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Orlando, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Baltimore, Maryland
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Rochester, Minnesota
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Las Vegas, Nevada
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Albany, New York
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., New York, New York
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Springfield, Oregon
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Charleston, South Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nashville, Tennessee
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bedford, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Dallas, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., McAllen, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., The Woodlands, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Webster, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Fairfax, Virginia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hampton, Virginia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Seattle, Washington
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Wenatchee, Washington
- Canada (6):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Edmonton, Alberta
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kelowna, British Columbia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Vancouver, British Columbia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., London, Ontario
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ottawa, Ontario
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Toronto, Ontario

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: https://vivli.org/

REFERENCES:
- [Derived] Petrylak DP, Tagawa ST, Kohli M, Eisen A, Canil C, Sridhar SS, Spira A, Yu EY, Burke JM, Shaffer D, Pan CX, Kim JJ, Aragon-Ching JB, Quinn DI, Vogelzang NJ, Tang S, Zhang H, Cavanaugh CT, Gao L, Kauh JS, Walgren RA, Chi KN. Docetaxel As Monotherapy or Combined With Ramucirumab or Icrucumab in Second-Line Treatment for Locally Advanced or Metastatic Urothelial Carcinoma: An Open-Label, Three-Arm, Randomized Controlled Phase II Trial. J Clin Oncol. 2016 May 1;34(13):1500-9. doi: 10.1200/JCO.2015.65.0218. Epub 2016 Feb 29. PMID 26926681

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants who died or discontinued treatment due to progressive disease (PD) were considered completers at the end of study. 8 participants were included in the "never treated" group due to death, PD, withdrawal, physician decision or protocol violation.
Groups:
- Docetaxel + Ramucirumab DP: Cycles repeat every 3 weeks until disease Progression, unacceptable toxicity, or withdrawal.
  Docetaxel: 75 mg/m2 on Day 1 of each 21-day cycle
  Ramucirumab (DP): 10 mg/kg IV on day 1 of each 21-day cycle
- Docetaxel + Icrucumab: Cycles repeat every 3 weeks until disease Progression, unacceptable toxicity, or withdrawal.
  Docetaxel: 75 mg/m2 on Day 1 of each 21-day cycle
  Icrucumab: 12 mg/kg IV on day 1 and Day 8 of each 21-day cycle
Period: Overall Study
Arm/Group | Docetaxel | Docetaxel + Ramucirumab DP | Docetaxel + Icrucumab
Started | 49 | 49 | 50
Received at Least 1 Dose of Study Drug | 45 | 46 | 49
Completed | 41 | 45 | 46
Not Completed | 8 | 4 | 4
Not completed — Lost to Follow-up | 1 | 0 | 0
Not completed — Withdrawal by Subject | 6 | 2 | 3
Not completed — Never Treated "Death" | 0 | 1 | 0
Not completed — Never Treated "PD" | 0 | 1 | 0
Not completed — Protocol Violation | 0 | 0 | 1
Not completed — Physician Decision | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All randomized participants who received at least 1 dose of study drug.
Groups:
- Docetaxel: Cycles repeat every 3 weeks until disease Progression, unacceptable toxicity, or withdrawal.
  Docetaxel: 75 mg/m2 on Day 1 of each 21-day cycle
- Total: Total of all reporting groups
Arm/Group | Docetaxel | Docetaxel + Ramucirumab DP | Docetaxel + Icrucumab | Total
Number analyzed (Participants) | 45 | 46 | 49 | 140
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.6 (11.45) | 66.7 (9.06) | 64.1 (10.38) | 65.7 (10.33)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 9 | 11 | 30
  Male | 35 | 37 | 38 | 110
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 3 | 2 | 9
  Not Hispanic or Latino | 41 | 43 | 47 | 131
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 5 | 2 | 4 | 11
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 2 | 0 | 2 | 4
  White | 36 | 43 | 42 | 121
  More than one race | 2 | 1 | 1 | 4
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Canada | 30 | 28 | 37 | 95
  United States | 15 | 18 | 12 | 45

OUTCOME MEASURES:

1. Primary Outcome: Progression-Free Survival (PFS)
Description: PFS time was the time from randomization until the date of objectively determined progressive disease (PD) or death due to any cause, whichever occurred first. According to Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST v1.1), PD was at least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study. In addition to the 20% relative increase, the sum must have also demonstrated an absolute increase of at least 5 millimeters (mm). The appearance of 1 or more new lesions and/or unequivocal progression of existing nontarget lesions was also considered progression. Participants without objectively determined PD who were alive at the end of the follow-up period (or lost to follow-up) were censored on the date of the participant's last complete radiographic tumor assessment; if no baseline or post-baseline radiologic assessment was available, the participant was censored at the date of randomization.
Time Frame: Randomization to Measured PD or Death From Any Cause (Up To 40 Months)
Population: All randomized participants who received at least one dose of study drug. Participants censored: docetaxel arm = 40; docetaxel and ramucirumab arm = 34; docetaxel and Icrucumab arm = 41.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Docetaxel | Docetaxel + Ramucirumab DP | Docetaxel + Icrucumab
Number analyzed (Participants) | 45 | 46 | 49
months | 2.8 [1.9 to 3.6] | 5.4 [3.1 to 6.9] | 1.6 [1.4 to 5.4]

2. Secondary Outcome: Percentage of Participants Achieving Objective Response Rate (ORR)
Description: Participants achieved an objective response if they had a best overall response of partial response (PR) or complete response (CR). According to RECIST v1.1, PR was defined as at least a 30% decrease in the sum of the diameters of target lesions (including the short axes of any target lymph node), taking as reference the baseline sum diameter; CR was the disappearance of all non-nodal target lesions, with the short axes of any target lymph node reduced to <10 mm, the disappearance of all nontarget lesions, and the normalization of tumor marker levels [if tumor markers were initially above the upper limit of normal (ULN)]. The percentage of participants who achieved an objective response=(number of participants with CR or PR)/(number of participants assessed)*100.
Time Frame: Randomization to Measured PD (Up to 40 Months)
Population: All randomized participants who received one dose of study drug.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Docetaxel: Cycles repeat every 3 weeks until disease Progression, unacceptable toxicity, or withdrawal.
  Docetaxel: Docetaxel: 75 mg/m2 on Day 1 of each 21-day cycle
Arm/Group | Docetaxel | Docetaxel + Ramucirumab DP | Docetaxel + Icrucumab
Number analyzed (Participants) | 45 | 46 | 49
percentage of participants | 8.9 [2.5 to 21.2] | 23.9 [12.6 to 38.8] | 12.2 [4.6 to 24.8]

3. Secondary Outcome: Duration of Response
Description: The duration of response was measured from the time measurement criteria were first met for a CR or PR (whichever was first recorded) until the first date of objectively documented progressive disease (taking as a reference for progressive disease the smallest measurement recorded since randomization) or the date of death, whichever occurred first. Data for participants who did not relapse or die were censored at the day of their last adequate tumor assessment. Duration of response was estimated by the Kaplan-Meier method.
Time Frame: First Criteria Met for CR or PR to Measured PD or Death From Any Cause (Up to 40 Months)
Population: All randomized participants received one dose of study drug and had CR or PR.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Docetaxel | Docetaxel + Ramucirumab DP | Docetaxel + Icrucumab
Number analyzed (Participants) | 4 | 11 | 6
months | 4.6 [2.6 to 5.6] | 4.6 [0.7 to 7.0] | NA [2.9 to NA] — The median and the upper limit was not estimable due to a small sample size and 2 participants had PD or Death.

4. Secondary Outcome: Number of Participants With Adverse Events (AEs)
Description: A summary of other nonserious AEs, and all SAE's, regardless of causality, is located in the Reported Adverse Events section.
Time Frame: Up To 41.7 Months
Population: All randomized participants who received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Docetaxel | Docetaxel + Ramucirumab DP | Docetaxel + Icrucumab
Number analyzed (Participants) | 45 | 46 | 49
Participants
  Any AE | 45 | 46 | 49
  Any SAE | 19 | 25 | 22

5. Secondary Outcome: Pharmacokinetics (PK) Maximum Concentration (Cmax) Ramucirumab
Time Frame: Cycle 1:Predose,1 hour(hr) post End of Infusion (EOI),48hr,72hr,168hr,336hr post-EOI;Cycle2:Predose,1hr post-EOI; Cycle3:Predose,1hr,48hr,72hr,168hr,336hr post-EOI; Cycle4:Predose,1hr post-EOI;Cycle6 and every other cycle thereafter:Predose,1hr Post EOI
Population: All randomized participants who received at least one dose of study drug and had evaluable PK data for Ramucirumab and there was no PK data for Docetaxel arm.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram/milliliter (ug/mL)
Groups:
- Docetaxel + Ramucirumab DP: Cycles repeat every 3 weeks until disease Progression, unacceptable toxicity, or withdrawal.
  Docetaxel: Docetaxel: 75 mg/m2 on Day 1 of each 21-day cycle
  Ramucirumab DP: Ramucirumab (DP): 10 mg/kg IV on day 1 of each 21-day cycle
Arm/Group | Docetaxel + Ramucirumab DP
Number analyzed (Participants) | 8
microgram/milliliter (ug/mL)
  Cycle 1 | 258 (27)
  Cycle 2: number analyzed (Participants) | 7
  Cycle 2 | 304 (31)
  Cycle 3: number analyzed (Participants) | 3
  Cycle 3 | 300 (13)
  Cycle 4: number analyzed (Participants) | 5
  Cycle 4 | 279 (40)
  Cycle 6: number analyzed (Participants) | 3
  Cycle 6 | 252 (57)

6. Secondary Outcome: PK: Minimum Concentration (Cmin) Ramucirumab
Time Frame: Cycle 2:Predose,1hr post-EOI;Cycle3:Predose,1hr,48hr,72hr,168hr,336hr, post-EOI;Cycle4:Predose,1hr post-EOI;Cycle6:Predose,1hr Post EOI
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram/milliliter (ug/mL)
Arm/Group | Docetaxel + Ramucirumab DP
Number analyzed (Participants) | 46
microgram/milliliter (ug/mL)
  Cycle 2: number analyzed (Participants) | 28
  Cycle 2 | 19.5 (56)
  Cycle 3: number analyzed (Participants) | 6
  Cycle 3 | 39.9 (34)
  Cycle 4: number analyzed (Participants) | 22
  Cycle 4 | 35.3 (60)
  Cycle 6: number analyzed (Participants) | 4
  Cycle 6 | 31.2 (61)

7. Secondary Outcome: PK: Cmax Icrucumab
Time Frame: Cycle 1:Predose,1 hr post-EOI, 48hr, 72hr Post-EOI; Cycle 3:Predose,EOI,1.5hr,24hr,48hr,72hr,168hr Post EOI
Population: All randomized participants who received at least one dose of study drug and had evaluable PK data for Icrucumab and there was no PK data for Docetaxel arm.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ug/mL
Arm/Group | Docetaxel + Icrucumab
Number analyzed (Participants) | 10
ug/mL
  Cycle 1 Cmax: number analyzed (Participants) | 8
  Cycle 1 Cmax | 474 (45)
  Cycle 3 Cmax: number analyzed (Participants) | 4
  Cycle 3 Cmax | 599 (27)

8. Secondary Outcome: PK: Cmin Icrucumab
Time Frame: Cycle 2:Predose,1hr post-EOI;Cycle 3:Predose,EOI,1.5hr,24hr,48hr,72hr,168hr Post EOI
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ug/mL
Arm/Group | Docetaxel + Icrucumab
Number analyzed (Participants) | 10
ug/mL
  Day 1 Cycle 2: number analyzed (Participants) | 1
  Day 1 Cycle 2 | NA (NA) — Geometric Mean and Geometric Coefficient of Variation was not calculable due to n=1.
  Day 1 Cycle 3: number analyzed (Participants) | 4
  Day 1 Cycle 3 | 153 (66)

9. Secondary Outcome: Number of Participants With Serum Anti-Ramucirumab Antibody Assessment
Description: Number of participants with at least one positive titer treatment emergent antibody positive neutralizing antibody detecting. A sample will be considered positive for anti-Ramucirumab antibodies if it exhibits a post-baseline antibody level exceeding the normal anti-Ramucirumab antibody level seen in healthy untreated individuals.
Time Frame: Cycle 1:Predose,EOI,1hr,48hr,72hr,168hr,336 hr post-EOI:Cycle 2:Predose,1hr post-EOI;Cycle 3:Predose,1hr,48hr,72hr,168hr,336hr post-EOI;Cycle 4:Predose,1hr post-EOI;Cycle 6:Predose,1hr post-EOI
Population: All randomized participants who received at least one dose of study drug and had baseline and post baseline anti-ramucirumab antibodies.
Measure: Count of Participants; unit: Participants
Arm/Group | Docetaxel + Ramucirumab DP
Number analyzed (Participants) | 43
Participants | 1

10. Secondary Outcome: Number of Participants With Serum Anti-Icrucumab Antibody Assessment
Description: A sample will be considered positive for anti-Icrucumab antibodies if it exhibits a post-baseline antibody level exceeding the normal anti-IMC-Icrucumab antibody level seen in healthy untreated individuals.
Time Frame: Cycle 1 Day 1 and Day 8 Predose and 1hr Post Dose
Population: Zero participants analyzed. Data not collected.
Groups:
- Docetaxel + Icrucumab: Cycles repeat every 3 weeks until disease Progression, unacceptable toxicity, or withdrawal.
  Docetaxel: Docetaxel: 75 mg/m2 on Day 1 of each 21-day cycle
  Icrucumab: 12 mg/kg IV on day 1 and Day 8 of each 21-day cycle
Arm/Group | Docetaxel + Icrucumab
Number analyzed (Participants) | 0

11. Secondary Outcome: Pharmacodynamics (PD): Change in Circulating Levels of Placental Growth Factor (PlGF)
Time Frame: 40 months
Population: Zero participants analyzed. Data not collected.
Arm/Group | Docetaxel | Docetaxel + Ramucirumab DP | Docetaxel + Icrucumab
Number analyzed (Participants) | 0 | 0 | 0

12. Secondary Outcome: PD: Change in Circulating Levels of Vascular Endothelial Growth Factor-A (VEGF-A)
Time Frame: 40 months
Population: Zero participants analyzed. Data not collected.
Arm/Group | Docetaxel | Docetaxel + Ramucirumab DP | Docetaxel + Icrucumab
Number analyzed (Participants) | 0 | 0 | 0

13. Secondary Outcome: PD: Change in Circulating Levels of Vascular Endothelial Growth Factor-B (VEGF-B)
Time Frame: 40 months
Population: Zero participants analyzed. Data not collected.
Arm/Group | Docetaxel | Docetaxel + Ramucirumab DP | Docetaxel + Icrucumab
Number analyzed (Participants) | 0 | 0 | 0

14. Secondary Outcome: PD: Change in Circulating Levels of Soluble Vascular Endothelial Growth Factor-1 (VEGFR-1)
Time Frame: 40 months
Population: Zero participants analyzed. Data not collected.
Arm/Group | Docetaxel | Docetaxel + Ramucirumab DP | Docetaxel + Icrucumab
Number analyzed (Participants) | 0 | 0 | 0

15. Secondary Outcome: PD: Change in Circulating Levels of Soluble Vascular Endothelial Growth Factor-2 (VEGFR-2)
Time Frame: 40 months
Population: Zero participants analyzed. Data not collected.
Arm/Group | Docetaxel | Docetaxel + Ramucirumab DP | Docetaxel + Icrucumab
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Description: All randomized participants who received at least one dose of study drug.
Arm/Group | Docetaxel | Docetaxel + Ramucirumab DP | Docetaxel + Icrucumab
Serious Adverse Events (participants affected / at risk) | 19/45 | 25/46 | 22/49
Other Adverse Events (participants affected / at risk) | 45/45 | 46/46 | 49/49
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Docetaxel (N=45) | Docetaxel + Ramucirumab DP (N=46) | Docetaxel + Icrucumab (N=49)
Anaemia (Blood and lymphatic system disorders) | 2 (2) | 1 (1) | 2 (2)
Febrile neutropenia (Blood and lymphatic system disorders) | 5 (6) | 9 (9) | 3 (3)
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 2 (3) | 4 (4) | 2 (2)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0) | 2 (2)
Cardio-respiratory arrest (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Left ventricular dysfunction (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Pericardial effusion (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1)
Ascites (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Duodenal perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Duodenal ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Gastric ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gastrointestinal ulcer haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Intestinal perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Large intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Mouth haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Oesophagitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pneumatosis intestinalis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Small intestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 3 (3) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Asthenia (General disorders) | 0 (0) | 1 (1) | 0 (0)
Device occlusion (General disorders) | 0 (0) | 1 (1) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0) | 0 (0)
Local swelling (General disorders) | 0 (0) | 0 (0) | 1 (1)
Multi-organ failure (General disorders) | 1 (1) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1) | 1 (1)
Pain (General disorders) | 0 (0) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 3 (3) | 0 (0)
Hepatic fibrosis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Arteritis infective (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Bronchopneumonia (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Escherichia bacteraemia (Infections and infestations) | 1 (2) | 0 (0) | 0 (0)
Eye infection staphylococcal (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Klebsiella sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Lobar pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Oral candidiasis (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 4 (4) | 1 (1)
Sepsis (Infections and infestations) | 2 (2) | 4 (4) | 0 (0)
Septic shock (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Stoma site infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 3 (3) | 3 (5)
Urosepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
White blood cell count decreased (Investigations) | 1 (2) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 2 (2) | 1 (1) | 2 (2)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hypovolaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Ischaemic stroke (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Paraesthesia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Spinal cord compression (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Haematuria (Renal and urinary disorders) | 2 (2) | 2 (2) | 1 (1)
Renal failure (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1)
Renal failure acute (Renal and urinary disorders) | 0 (0) | 2 (2) | 1 (1)
Renal tubular necrosis (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Urinary tract obstruction (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 2 (2)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 2 (2)
Swelling face (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Accelerated hypertension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Circulatory collapse (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 2 (2)
Hypotension (Vascular disorders) | 1 (1) | 0 (0) | 1 (1)
Phlebitis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Docetaxel (N=45) | Docetaxel + Ramucirumab DP (N=46) | Docetaxel + Icrucumab (N=49)
Anaemia (Blood and lymphatic system disorders) | 10 (14) | 11 (44) | 20 (49)
Leukopenia (Blood and lymphatic system disorders) | 2 (3) | 2 (2) | 5 (14)
Neutropenia (Blood and lymphatic system disorders) | 11 (18) | 9 (15) | 13 (25)
Thrombocytopenia (Blood and lymphatic system disorders) | 4 (8) | 8 (23) | 3 (4)
Tachycardia (Cardiac disorders) | 3 (4) | 1 (1) | 1 (1)
Lacrimation increased (Eye disorders) | 3 (3) | 12 (18) | 5 (5)
Vision blurred (Eye disorders) | 2 (2) | 2 (2) | 4 (5)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1) | 3 (3) | 1 (3)
Abdominal pain (Gastrointestinal disorders) | 5 (5) | 10 (11) | 6 (6)
Abdominal pain lower (Gastrointestinal disorders) | 2 (2) | 3 (4) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 2 (2) | 3 (4) | 1 (3)
Constipation (Gastrointestinal disorders) | 9 (14) | 9 (12) | 15 (17)
Diarrhoea (Gastrointestinal disorders) | 11 (16) | 25 (44) | 22 (30)
Dry mouth (Gastrointestinal disorders) | 3 (5) | 4 (4) | 5 (6)
Dyspepsia (Gastrointestinal disorders) | 3 (4) | 3 (4) | 3 (3)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 5 (6) | 1 (2)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 1 (1) | 3 (4)
Nausea (Gastrointestinal disorders) | 12 (19) | 24 (36) | 24 (40)
Oral pain (Gastrointestinal disorders) | 0 (0) | 3 (3) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 7 (10) | 15 (29) | 4 (4)
Vomiting (Gastrointestinal disorders) | 7 (7) | 14 (20) | 14 (21)
Asthenia (General disorders) | 2 (3) | 6 (7) | 3 (4)
Chills (General disorders) | 5 (5) | 7 (8) | 2 (3)
Fatigue (General disorders) | 36 (63) | 38 (108) | 38 (135)
Influenza like illness (General disorders) | 4 (5) | 2 (2) | 3 (3)
Mucosal inflammation (General disorders) | 4 (4) | 10 (19) | 3 (9)
Non-cardiac chest pain (General disorders) | 1 (1) | 5 (5) | 1 (1)
Oedema peripheral (General disorders) | 9 (10) | 17 (27) | 24 (49)
Pain (General disorders) | 1 (1) | 2 (5) | 3 (4)
Peripheral swelling (General disorders) | 2 (2) | 1 (1) | 5 (5)
Pyrexia (General disorders) | 5 (6) | 11 (14) | 11 (15)
Candida infection (Infections and infestations) | 4 (4) | 3 (4) | 2 (3)
Oral candidiasis (Infections and infestations) | 3 (4) | 3 (3) | 1 (1)
Pneumonia (Infections and infestations) | 3 (3) | 4 (4) | 1 (1)
Rhinitis (Infections and infestations) | 2 (2) | 3 (3) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 2 (2) | 3 (4)
Urinary tract infection (Infections and infestations) | 9 (10) | 9 (12) | 6 (9)
Fall (Injury, poisoning and procedural complications) | 3 (3) | 1 (1) | 1 (2)
Infusion related reaction (Injury, poisoning and procedural complications) | 2 (2) | 1 (1) | 6 (10)
Blood creatinine increased (Investigations) | 5 (7) | 3 (3) | 4 (8)
Neutrophil count decreased (Investigations) | 7 (15) | 6 (7) | 7 (20)
Weight decreased (Investigations) | 1 (1) | 7 (10) | 3 (4)
Weight increased (Investigations) | 0 (0) | 1 (2) | 5 (5)
White blood cell count decreased (Investigations) | 6 (6) | 1 (2) | 3 (4)
Decreased appetite (Metabolism and nutrition disorders) | 19 (30) | 26 (39) | 25 (41)
Dehydration (Metabolism and nutrition disorders) | 6 (6) | 9 (14) | 10 (19)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 3 (3) | 2 (2) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 2 (2) | 4 (5)
Hypomagnesaemia (Metabolism and nutrition disorders) | 3 (4) | 2 (2) | 3 (4)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 3 (7)
Arthralgia (Musculoskeletal and connective tissue disorders) | 11 (20) | 11 (17) | 12 (17)
Back pain (Musculoskeletal and connective tissue disorders) | 7 (8) | 6 (10) | 7 (9)
Bone pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 5 (9) | 1 (1)
Flank pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 3 (3) | 2 (4)
Groin pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0) | 2 (2)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 4 (4) | 8 (19) | 7 (10)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3) | 3 (5)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (3) | 4 (5)
Myalgia (Musculoskeletal and connective tissue disorders) | 6 (8) | 12 (30) | 7 (11)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2) | 7 (11) | 7 (10)
Dizziness (Nervous system disorders) | 3 (6) | 8 (12) | 10 (11)
Dysgeusia (Nervous system disorders) | 17 (25) | 14 (26) | 16 (32)
Headache (Nervous system disorders) | 3 (5) | 9 (13) | 6 (6)
Hypoaesthesia (Nervous system disorders) | 1 (1) | 3 (3) | 2 (3)
Neuropathy peripheral (Nervous system disorders) | 6 (6) | 11 (21) | 8 (14)
Paraesthesia (Nervous system disorders) | 6 (6) | 7 (8) | 4 (5)
Peripheral sensory neuropathy (Nervous system disorders) | 6 (11) | 7 (8) | 6 (8)
Anxiety (Psychiatric disorders) | 2 (2) | 1 (1) | 4 (4)
Depression (Psychiatric disorders) | 0 (0) | 5 (5) | 2 (2)
Insomnia (Psychiatric disorders) | 4 (4) | 10 (16) | 17 (26)
Haematuria (Renal and urinary disorders) | 2 (4) | 15 (37) | 4 (7)
Hydronephrosis (Renal and urinary disorders) | 0 (0) | 4 (4) | 1 (1)
Proteinuria (Renal and urinary disorders) | 1 (5) | 3 (4) | 5 (6)
Urinary retention (Renal and urinary disorders) | 2 (2) | 4 (6) | 1 (1)
Scrotal oedema (Reproductive system and breast disorders) | 1/35 (1) | 3/37 (4) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (8) | 18 (23) | 16 (19)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 11 (14) | 12 (16) | 16 (25)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 4 (5) | 5 (8)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 20 (23) | 0 (0)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 3 (3) | 2 (3)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 6 (7) | 3 (4)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 10 (11) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 5 (7) | 3 (4)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 3 (3)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 5 (5) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 22 (28) | 27 (34) | 26 (30)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 3 (3) | 2 (3) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 5 (7) | 2 (2)
Ecchymosis (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (4) | 1 (1)
Nail discolouration (Skin and subcutaneous tissue disorders) | 3 (3) | 5 (5) | 1 (1)
Nail disorder (Skin and subcutaneous tissue disorders) | 4 (4) | 2 (2) | 1 (1)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 1 (1) | 4 (5) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 3 (4) | 1 (1) | 1 (2)
Rash (Skin and subcutaneous tissue disorders) | 2 (2) | 3 (4) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 8 (12) | 3 (5) | 4 (6)
Flushing (Vascular disorders) | 1 (1) | 3 (4) | 5 (5)
Hypertension (Vascular disorders) | 3 (8) | 10 (15) | 1 (1)
Hypotension (Vascular disorders) | 5 (8) | 8 (8) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days